

## Post Marketing Surveillance Study -Retrospective Study Endofast Reliant SCP Protocol

| Document No. | Revision | Page |
|--------------|----------|--------|
| CL-SCP-60-04 | 00 | 1 of 2 |



## Post Marketing Clinical Follow Up (PMCF) Study

A Retrospective Study for collecting data on the Safety and Performance of the EndoFast Reliant SCP in Vaginal Wall Reinforcement Study Protocol

March 13, 2017



## Post Marketing Surveillance Study -Retrospective Study Endofast Reliant SCP Protocol

| Document No. | Revision | Page |
|--------------|----------|--------|
| CL-SCP-60-04 | 00 | 2 of 2 |

## **Study Synopsis**

| Study Design | A Single arm, single site, retrospective cohort Post Marketing Surveillance Study Evaluating the Safety and |
|---|---|
| | Performance of the <i>EndoFast Reliant SCP</i> for apical support |
| Study device: | EndoFast Reliant SCP |
| Intended use: | The <i>EndoFast Reliant SCP</i> is indicated for fixation of surgical mesh to tissue for tissue reinforcement during laparotomy or laparoscopic Sacrocolpopexy approach. |
| Device Regulatory status: | CE, AMAR and FDA Approval |
| Objective: | The objective of this study is to collect data on the anatomical cure and safety of the EndoFast Reliant SCP |
| Medical Centers | One site in Germany Catholic Hospital Hoxter, Germany Dr. Bettin |
| Population: | Female subjects >18 years old that underwent Pelvic Organ Prolapse repair utilizing the EndoFast Reliant SCP |
| Procedure: | Pelvic Organ Prolapse repair utilizing the EndoFast Reliant SCP |
| Follow-up: | Upon availability of the data (retrospective study) |
| Safety Endpoint: | The safety endpoint counts the rate of peri and post-<br>operative device related Adverse Events. |
| Effectiveness Endpoints: | measures the relative improvement in Pelvic Organ Prolapse staging using the POPQ grading system |
| Inclusion criteria | All Female subjects >18 years old that underwent Pelvic Organ Prolapse repair utilizing the EndoFast Reliant SCP |
| Exclusion criteria | Patients without follow-up |
| Sponsor: | IBI, Israel Biomedical Innovations Ltd. |
| | 2 Ha-Eshel St., P.O.BOX 3081, Caesarea Industrial Park, |
| | 3088900 - Israel |
| | Tel: +972-4-6277166 |
| | Fax: +972-4-6277266 |